CLINICAL TRIAL: NCT00053820
Title: A Randomized Controlled Trial of Interferon-alpha, Interleukin-2 and 5-Fluorouracil vs. Interferon-alpha Alone in Patients With Advanced Renal Cell Carcinoma
Brief Title: Interferon Alfa With or Without Interleukin-2 and Fluorouracil in Treating Patients With Advanced Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269480; MRC-RE04; EORTC-30012; EU-20231; ISRCTN46518965
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-08

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha; Fluorouracil

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Drug: fluorouracil

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining interferon alfa with interleukin-2 and fluorouracil may kill more tumor cells. It is not yet known whether interferon alfa is more effective with or without interleukin-2 and fluorouracil in treating metastatic kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa combined with interleukin-2 and fluorouracil to that of interferon alfa alone in treating patients who have advanced metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression-free and overall survival of patients with advanced metastatic renal carcinoma treated with interferon alfa with or without interleukin-2 and fluorouracil.
* Compare the toxicity of these regimens in these patients.
* Assess the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (Interferon alfa monotherapy): Patients receive interferon alfa subcutaneously (SC) on days 1, 3, and 5. Treatment continues weekly for at least 9 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II (Interferon alfa, interleukin-2, and fluorouracil combination therapy): Patients receive interferon alfa SC on day 1 of weeks 1 and 4 and days 1, 3, and 5 of weeks 2, 3, 5, 6, 7, and 8. Patients also receive interleukin-2 SC twice daily on days 3-5 of weeks 1 and 4 and once daily on days 1, 3, and 5 of weeks 2 and 3. Patients then receive fluorouracil IV on day 1 of weeks 5-8. Treatment repeats every 10 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at 9, 19, and 26 weeks, and then at 8 months.

Patients are followed at 8, 10, and 12 months, every 4 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 670 patients (335 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Advanced metastatic disease that requires treatment
* Measurable disease (single bone lesions not included)
* No brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 to 81

Performance status

* WHO 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No myocardial infarction within the past 6 months
* No unstable angina pectoris

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 6 months after study participation
* No other concurrent disease or prior malignancy that would preclude study treatments or comparisons
* No concurrent active infection requiring antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior endocrine therapy
* No concurrent corticosteroids

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Prior resection of the primary tumor recommended but not required
* No prior major organ allografts

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2002-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Time to progression as measured by RECIST criteria
Comparison of toxicity levels (Grade III and IV)
Comparison of quality of life before, during, after completion of study treatment
Impact of the treatment regimens on health economics

CONTACTS AND LOCATIONS:
Overall Officials: Martin E. Gore, MD — Royal Marsden NHS Foundation Trust; Peter F.A. Mulders, MD, PhD — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (12):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Klinikum Kassel, Kassel, Germany
- Netherlands (5):
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
- National Cancer Institute - Bratislava, Bratislava, Slovakia

REFERENCES:
- [Result] Gore ME, Griffin CL, Hancock B, Patel PM, Pyle L, Aitchison M, James N, Oliver RT, Mardiak J, Hussain T, Sylvester R, Parmar MK, Royston P, Mulders PF. Interferon alfa-2a versus combination therapy with interferon alfa-2a, interleukin-2, and fluorouracil in patients with untreated metastatic renal cell carcinoma (MRC RE04/EORTC GU 30012): an open-label randomised trial. Lancet. 2010 Feb 20;375(9715):641-8. doi: 10.1016/S0140-6736(09)61921-8. Epub 2010 Feb 10. PMID 20153039
- [Result] Gore ME: Interferon-α (IFN), interleukin-2 (IL2) and 5-fluorouracil (5FU) vs IFN alone in patients with metastatic renal cell carcinoma (mRCC): results of the randomised MRC/EORTC RE04 trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-5039, 2008.